CLINICAL TRIAL: NCT00478764
Title: Intracameral Use of Triamcinolone and Gatifloxacin Versus Standard Postoperative Steroid and Antibiotic Eye Drops After Cataract Surgery
Brief Title: Intraocular Steroid After Cataract Surgery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dean Health System (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOSS
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Cataract
Keywords: intraocular; triamcinolone; gatifloxicin; inflammation; visual acuity
MeSH Terms: conditions — Cataract; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: intraocular triamcinolone and gatifloxicin

SUMMARY:
The use of one dose of an antibiotic and steroid injected into the eye at the end of cataract surgery is as safe and effective as the post operative use of eyedrops after cataract surgery.

DETAILED DESCRIPTION:
This prospective randomized controlled trial included 80 eyes of 40 patients having routine phacoemulsification of cataract. Patients between 40 and 80 years of age who met enrollment criteria, required cataract surgery in both eyes, and agreed to participate, were enrolled in the study over a nine month period in 2006 at the office of one cataract surgeon. Eyes were randomly assigned to receive either the eye drop or injection protocol on the initial consultative visit. All surgery was preformed by one surgeon (JGS) using topical anesthesia, the Infiniti phacoemulsification system (Alcon) and an Acrysof SN60WF (Alcon) intraocular lens. The fellow eye was operated upon using the same technique and instrumentation two weeks later and was assigned to the group opposite the first eye. All eyes were examined by the operating surgeon at days 1, 8, 15, 30 and 90 postoperatively with uncorrected visual acuity, best corrected visual acuity, intraocular pressure, corneal edema, anterior chamber cell and flare recorded.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients to enter the study included age 40 to 80 years, clinically significant cataract in both eyes, the patient's willingness to enter the study and have cataract surgery preformed on each eye in a sequentially within a two or three week time frame.

Exclusion Criteria:

* Exclusion criteria included a history of glaucoma, retinopathy of any type, pseudoexfoliation, other significant ocular co morbidity and systemic diabetes.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
visual acuity | 90 days

SECONDARY OUTCOMES:
intraocular inflammation | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan G Stock, MD, Principal Investigator — Dean Health Systems
Locations (1):
- Davis Duehr Dean Baraboo, Baraboo, Wisconsin, United States

REFERENCES:
- [Background] Gills JP, Gills P. Effect of intracameral triamcinolone to control inflammation following cataract surgery. J Cataract Refract Surg. 2005 Aug;31(8):1670-1. doi: 10.1016/j.jcrs.2005.07.023. No abstract available. PMID 16129313